CLINICAL TRIAL: NCT02512848
Title: The Feasibility Study of Li Brush for the Screening of Endometrial Cancer in the Postmenopausal Period
Brief Title: The Feasibility Study of the Li Brush for the Screening of Endometrial Cancer in the Postmenopausal Period
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AHCR2014-007
Record Dates: First submitted 2015-07-08; First posted 2015-07-31 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Endometrial Neoplasms
Keywords: postmenopause; endometrial sampling; vaginal bleeding
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — endometrial sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- endometrial neoplasms: patients with risk of endometrial cancer in the postmenopausal period

SUMMARY:
Investigators aim to collect endometrial sampling with Li Brush among target population who have risks for endometrial neoplasm, then Fractional curettage should performed with these participants, investigators intend to compare the pathological diagnosis results of cytology and fractional curettage to evaluate the sensitivity of Li Brush and investigators expect that the brush can be used for screening of endometrial cancer in the postmenopausal period in the clinic.

DETAILED DESCRIPTION:
Investigators screen the suitable participants according to the inclusion and exclusion standards, and then collect their endometrial sampling with Li Brush. Pathologists will help to decide the cytology obtained by Li Brush and histology diagnosis of the endometrial sampling. Comparing the pathological diagnosis results of cytology and histology, investigators want to prove the feasibility of cytology diagnosis of endometrial cancer in the postmenopausal period, as the same time, investigators intend to evaluate the possible factors that affecting the precision of Li Brush for endometrial cancer in the postmenopausal period.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal abnormal uterine bleeding;
2. Ultrasound of the pelvic showed thickened endometrial ( usually more than 5mm) ;
3. Family history of endometrial cancers;
4. Other participants with risks for endometrial cancer (such as fat, Lynch Syndrome and so on)

Exclusion Criteria:

1. Cervical cancer;
2. Fever (body's temperature is higher than 37.5 degrees );
3. Vaginitis (excluding atrophic vaginitis);
4. Patients who cannot bear the operation;
5. Coagulation disorders;
6. Pregnancy and suspected pregnancy.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants with risks of endometrial cancer in the postmenopausal period
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Compare the new diagnosis method with gold standard via Kappa statistic | one week within the enrollment
  Kappa statistic will be used to access the agreement of the two diagnosis results. The diagnosis result is dichotomous data: having endometrial cancer or not. The safety risk is the same as it of the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Qiling Li, MD, PHD, Principal Investigator — The First Affliated Hospital of Xi'an Jiaotong University
Locations (1):
- The First Affliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meads C, Sutton A, Malysiak S, Kowalska M, Zapalska A, Rogozinska E, Baldwin P, Rosenthal A, Ganesan R, Borowiack E, Barton P, Roberts T, Sundar S, Khan K. Sentinel lymph node status in vulval cancer: systematic reviews of test accuracy and decision-analytic model-based economic evaluation. Health Technol Assess. 2013 Dec;17(60):1-216. doi: 10.3310/hta17600. PMID 24331128
- [Background] Demirkiran F, Yavuz E, Erenel H, Bese T, Arvas M, Sanioglu C. Which is the best technique for endometrial sampling? Aspiration (pipelle) versus dilatation and curettage (D&C). Arch Gynecol Obstet. 2012 Nov;286(5):1277-82. doi: 10.1007/s00404-012-2438-8. Epub 2012 Jul 6. PMID 22766754
- [Background] Kipp BR, Medeiros F, Campion MB, Distad TJ, Peterson LM, Keeney GL, Halling KC, Clayton AC. Direct uterine sampling with the Tao brush sampler using a liquid-based preparation method for the detection of endometrial cancer and atypical hyperplasia: a feasibility study. Cancer. 2008 Aug 25;114(4):228-35. doi: 10.1002/cncr.23636. PMID 18548528
- [Background] Williams AR, Brechin S, Porter AJ, Warner P, Critchley HO. Factors affecting adequacy of Pipelle and Tao Brush endometrial sampling. BJOG. 2008 Jul;115(8):1028-36. doi: 10.1111/j.1471-0528.2008.01773.x. PMID 18651884